CLINICAL TRIAL: NCT06182241
Title: Identifying and Addressing Barriers to Retention in the Cervical Cancer Treatment Cascade Among Women With HIV in South Africa: Part 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amelia M. Stanton, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7356E
Record Dates: First submitted 2023-11-30; First posted 2023-12-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer; Hiv
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant intervention (Experimental): The intervention group will likely consist of one to two sessions, conducted in-person, coupled with text- or phone-based client navigation.The intervention group will complete three major assessments: baseline (T1), at the conclusion of the intervention (T2), and a three-month follow-up (T3). Until the follow-up assessment, the interventionist will send participants up to 6 SMS messages (one-way) per month. The content of these messages will be developed collaboratively between the participant and the interventionist during the second session; messages could include reminders about follow-ups and/or prompts to use new skills and resources for navigating specific barriers.
  Interventions: Behavioral: Retention in cervical cancer care intervention
- Treatment as usual (No Intervention): The treatment as usual (TAU) group will receive treatment as usual, including being notified of their abnormal Pap results via SMS and instructed to set up a follow-up appointment, as is typical in routine care. The TAU group will complete the T1 assessment and will complete T2 assessment two-months post-baseline.

INTERVENTIONS:
Behavioral: Retention in cervical cancer care intervention — Aim 1 data will inform this intervention, however the participant intervention will likely be one or two sessions, conducted in-person, coupled with text- or phone-based client navigation with women who received abnormal high-risk Pap smear results. We anticipate that the intervention may integrate (1) information to improve awareness of cervical cancer susceptibility and treatment, (2) motivational interviewing to assess pros and cons of attending a follow-up appointment and completing treatment; (3) brief cognitive behavioral therapy (CBT) skills to reduce individual-level barriers, (4) problem-solving to increase social support, and (5) patient navigation tools to mitigate clinic-level challenges.
  Arms: Participant intervention

SUMMARY:
The investigators will conduct the formative work that is necessary to develop a novel, multi-level intervention (inclusive of patient- and provider-level components), which will increase awareness of and modify the complex, intersecting factors that contribute to cervical cancer development among cisgender women with HIV (WWH). In Aim 1a, the investigators will explore the multi-level barriers and facilitators to follow-up appointment attendance among WWH who have had a recent high-risk abnormal Pap smear in the past six months, via qualitative interviews with WWH who have either attended at least one follow-up visit (n<10) or have not yet attended a follow-up visit (n<10). In Aim 1b, the investigators will explore provider awareness of the HIV-cervical cancer relationship and perspectives on barriers to retention in care via qualitative interviews (n<8). For Aim 2, The study team will leverage the Aim 1 data, develop a patient-level intervention (1-2 sessions) and a provider toolkit, with the goal of increasing retention in care among WWH who are at heightened risk for cervical cancer. The study team will seek feedback on the manual and the toolkit from providers and from a community advisory board. In Aim 3a, the investigators will test the feasibility and acceptability of the intervention in a pilot randomized control trial (RCT) (n<60). The study team will also assess (1) changes in self-efficacy to attend cervical cancer-related healthcare appointments pre-post intervention, (2) the proportion of women who attend a follow-up appointment, and, of those participants, (3) the proportion of women who complete the next phase of treatment. In Aim 3b, the investigators will explore the feasibility of intervention implementation in the clinic and acceptability of the provider-level intervention components in qualitative interviews with providers, clinic staff, the interventionalists, and other key stakeholders (n<10).

ELIGIBILITY:
Inclusion Criteria:

* Having a cervix
* Aged 18+
* Living with HIV
* Recent high-risk abnormal Pap results within the last month (if needed, we may increase the range by up to 6 months to ensure that we meet our targets).

Exclusion Criteria:

* Younger than 18 years old
* HIV-negative
* No cervix/history of hysterectomy
* Recent normal or low-risk abnormal Pap results
* Unable to provide informed consent or assent in English or isiZulu and/or have a significant psychiatric illness (e.g., active psychotic disorder or untreated bipolar disorder) that could interfere with participation will be excluded. Potential participants will also be asked if they have any health conditions that make it difficult for them to travel to the clinic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | About 1-2 months after the start of intervention and at about 4 months after the start of the intervention
  Feasibility will be demonstrated if all three are met by participants: (1) 50% of participants who are approached choose to enroll; (2) 70% of participants complete the intervention; and (3) 60% complete the 3-month follow-up. Feasibility of the implementation of the intervention will be explored in interviews with providers, clinic staff, interventionalists, and other relevant stakeholders.
Acceptability of the intervention | About 1-2 months after the start of intervention and at about 4 months after the start of the intervention
  Acceptability will be measured using the seven component constructs of the acceptability of health care interventions framework using a five-point Likert style scale. The seven components include affective attitude (i.e., how an individual feels about the intervention), burden, ethicality (i.e., the extent to which the intervention aligns with one's value system), intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy. Acceptability will be demonstrated if, on average, at least 75% of the participants rate five or more of the items on the eight-item Acceptability of Healthcare Interventions Questionnaire with a 4 or a 5 on the Likert-style scale. Acceptability of the intervention will also be explored in interviews with providers, clinic staff, interventionalists, and other relevant stakeholders.

SECONDARY OUTCOMES:
Self-efficacy to attend cervical cancer-related health care appointment | Start of the intervention and about 1-2 months after the start of intervention
  This will be measured by comparing change scores from baseline to post-intervention between the intervention and TAU groups.
Follow-up appointment attendance | About 4 months after the start of the intervention
  This will be measured by comparing the proportions between intervention and TAU groups.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
- MatCH Research Unit (MRU), a Division of the Wits Health Consortium, University of Witwatersrand, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No